CLINICAL TRIAL: NCT07166939
Title: A Phase 4, Multicenter, Cluster Randomized, Open-label, Intervention Versus Usual Care, Controlled Study on the Effect of Emergency Department Initiation of Airsupra on Asthma Outcomes
Brief Title: 45th Multicenter Airway Research Collaboration
Acronym: MARC-45
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Carlos A. Camargo, Jr., Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025P002364
Record Dates: First submitted 2025-09-09; First posted 2025-09-11 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Asthma Acute; Asthma Exacerbation; Asthma; Asthma Control Level
Keywords: asthma; emergency department; airsupra; randomized trial; acute asthma recurrence; acute asthma relapse; asthma control; acute asthma; asthma exacerbation
MeSH Terms: conditions — Asthma; Emergencies

STUDY DESIGN:
Intervention Model Description: cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): usual care
- Intervention (Active Comparator): Airsupra PRN
  Interventions: Drug: Airsupra

INTERVENTIONS:
Drug: Airsupra — 1 dose (2 inhalations) PRN, with maximum of 6 doses (12 inhalations) in a 24-hour period
  Arms: Intervention

SUMMARY:
The study is a randomized controlled trial on the effect of emergency department initiation of Airsupra on acute asthma "recurrence" at 3 months and other related outcomes (acute asthma relapse, asthma control).

DETAILED DESCRIPTION:
Acute asthma (or asthma exacerbation) is common and costly. In the USA, acute asthma accounts for approximately 2 million emergency department (ED) visits per year; approximately 10-20% of patients are admitted and, among those discharged, approximately 15-20% relapse (i.e., return to the ED for further treatment of their index exacerbation). A 2000 Cochrane review evaluated if starting inhaled corticosteroids (ICS) at ED discharge would lower risk of relapse during the 2-3 weeks after the ED visit. The meta-analysis included three randomized controlled trials (RCTs) and found borderline significant evidence that ICS initiation lowered risk of relapse during the 2-3 weeks after ED discharge (total n=909 patients; OR 0.68; 95%CI 0.46-1.02).

For decades, asthma experts have tried to increase ED-based prescribing of ICS to ED patients with asthma but uptake has been slow. In addition to reluctance among ED clinicians to prescribe a "lifelong" medication, a challenge has been patients' perception that they do not receive any immediate symptom relief from the new (ICS only) inhaler - i.e., "it does not work as well" as their regular (albuterol) inhaler. FDA approval of Airsupra (with both albuterol and budesonide in one inhaler) provides a unique opportunity to introduce ICS (along with albuterol) to ED patients with acute asthma.

The proposed trial is a cluster randomized, open-label, intervention vs usual care, controlled study on the effect of ED initiation of Airsupra on acute asthma recurrence at 3 months (primary outcome) - i.e., a combination of acute asthma "relapse" (by 3 weeks) plus subsequent exacerbations. The trial is powered to assess a 33% reduction in recurrence at 3 months and will have ample power to explore asthma control, both overall and in important subgroups (e.g., stratified by age, sex, race/ethnicity, BMI, current asthma medications, and number of ED visits for acute asthma in the past year). Randomization of sites will be stratified by US region to increase likelihood that the two groups are similar at baseline.

Patients will be enrolled by members of the Multicenter Asthma Research Collaboration (MARC), within the Emergency Medicine Network (EMNet). This research network was founded in 1996 with the original goal of performing clinical research on acute asthma. Massachusetts General Hospital is the EMNet Coordinating Center and will not participate in patient enrollment. Patient inclusion criteria include: acute asthma (i.e., fulfill American Thoracic Society criteria for asthma; age 18-54 years (to minimize contamination by COPD and to permit testing of effect modification by age); decision by ED attending to discharge patient to home on short course of systemic corticosteroids (to "validate" that patient truly had an asthma exacerbation); and informed consent. Patient exclusion criteria include: prior diagnosis of COPD, use of systemic corticosteroids in the past 2 weeks (to avoid enrollment of severe persistent asthma or patients presenting to ED with an acute asthma relapse, rather than their index presentation of acute asthma); comorbid complications (e.g., concurrent pneumonia, influenza, COVID-19); lack of a working cell phone and working email address (having both is common today and will increase follow-up rates); expected lack of availability for text and/or telephone follow-up at approximately 3, 6, and 12 weeks after the ED visit; or prior enrollment in this study.

All patients will undergo a short, structured interview in the ED and a focused ED chart review, using previously developed instruments for ED-based asthma research. Site investigators will enter these data into a REDCap database created and managed at the EMNet Coordinating Center in Boston. Based on their random site assignment (intervention vs usual care), intervention sites will put enrolled patients on a short course of systemic corticosteroids (e.g., prednisone 50 mg daily x 5 days) and Airsupra PRN (rescue inhaler). Usual care sites will manage patients per usual care. All patients will receive a brief educational handout about asthma.

At approximately 3, 6, and 12 weeks after the ED discharge, EMNet staff will follow-up with patients about their clinical course (including acute asthma relapse, asthma control, medication use), and potential adverse effects from any of the medications prescribed at ED discharge. Most follow-up assessments will be by telephone interview, but texts will be used per patient preference and/or to increase completeness of follow-up. Asthma control will be assessed using the AirQ, a 10-item instrument. EMNet staff will enter data into the REDCap database.

Patients will sign medical release forms so that EMNet staff in Boston can collect medical records for the 12 months before enrollment and the first 3 months after enrollment. These records will come from the enrolling hospital or hospital system/network, along with the patient's primary care provider and, when applicable, their asthma specialist (allergist/immunologist, pulmonologist, asthma center). EMNet staff will review these medical records to identify repeat asthma exacerbations (ie, recurrence) and the patient's current medications at the end of the 3-month follow-up period. EMNet staff will enter data into the REDCap database.

The primary outcome is acute asthma "recurrence" (i.e., any urgent or unscheduled visit to a clinician for worsening asthma symptoms) during the 3 months after the ED visit. This outcome differs from acute asthma "relapse" which is typically assessed during the 3 weeks after the ED visit; prior research indicates that symptoms of an exacerbation typically resolve by 1-2 weeks while biochemical evidence of the exacerbation resolves by 3 weeks. The frequency of recurrence in this unique, ED-based population is not known - but the investigators' best estimate for the usual care group is approximately 33% (i.e., they will experience 15% relapse in the first 3 weeks then additional events during the 9 weeks of fall/winter that follow.) The main secondary outcome will be asthma control at 3 months after the ED visit. Other secondary outcomes include acute asthma relapse (3 weeks) and post-ED initiation of Airsupra (any time during follow-up).

Data analysis will describe patient characteristics, overall and in the two randomly allocated groups (15 intervention sites, 15 usual care sites). The primary outcome (acute asthma recurrence at 3 months after the index ED visit) will be analyzed using time-to-event data, in both unadjusted and multivariable models. Covariates will be major sociodemographic factors (e.g., age, sex, race/ethnicity, insurance) and clinical factors with an observed association (P<0.20) with the recurrence outcome. The main secondary outcome (3-month asthma control) will be compared using t-test or Mann-Whitney U-test, as appropriate. Repeated measures are not necessary since the investigators will focus on 3-month asthma control; asthma control at baseline is non-interpretable in the context of the index exacerbation. The investigators will not do an interim analysis given the short study enrollment (September to December 2025), across 30 centers, and given the demonstrated safety of Airsupra (per FDA approval).

Power calculations, based on acute asthma recurrence at 3 months (with an estimated intra-cluster correlation [ICC] of 0.02), suggest that 1290 patients are needed to detect a 33% reduction in recurrence (e.g., 22% recurrence in the Airsupra group vs. 33% recurrence in the usual care group). The main secondary outcome, asthma control, will require fewer patients. The investigators anticipate 70% follow-up of enrolled patients at 3 months and, therefore, have increased the target sample size to 1860 total patients (930 per arm; 62 per site). Based on experience with ED-based asthma research since the 1990s, the investigators believe that each site, over 4 months (September to December 2025), can enroll at least 62 adult patients with acute asthma. (30 sites x 62 patients/site = 1860)

ELIGIBILITY:
INCLUSION CRITERIA:

* acute asthma
* age 18.0 to 54.9 years
* English and/or Spanish speaking
* decision by ED attending to discharge patient to home on short course of systemic corticosteroids
* (intervention group only) Willingness to use Airsupra as their rescue inhaler for next 3 months
* demonstration of acceptable MDI administration technique
* provision of informed consent prior to any study-specific procedures

EXCLUSION CRITERIA:

* involvement in the planning and/or conduct of the study
* previous enrolment in the present study
* prior diagnosis of COPD, chronic bronchitis, or emphysema
* use of systemic corticosteroids in the past 2 weeks
* participation in another clinical study with an investigational product during the past 4 weeks or the 3 months after enrollment in the current study
* concurrent pneumonia, influenza, or COVID-19
* clinically significant cardiovascular disease or clinically significant cancer
* patients with known hypersensitivity to Airsupra, albuterol sulfate, budesonide, or any of the excipients of the product
* (for women only, by self-report):
* currently pregnant
* currently breastfeeding,
* (among sexually active women of child-bearing age only) not using adequate contraception over the last 3 months, or no plan to use adequate contraception over the next 3 months
* lack of a working cell phone and working email address
* expected lack of availability for text and/or telephone follow-up at approximately 3, 6, and 12 weeks after the ED visit
* inability to provide an alternate contact with a working cell phone and working email address.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1860 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
acute asthma recurrence | 3 months
  any urgent or unscheduled visit to a clinician for worsening asthma symptoms during the 3 months after the index ED visit

SECONDARY OUTCOMES:
asthma control | 3 months
  asthma control at 3 months after the index ED visit, as measured by AIRQ
acute asthma relapse | 3 weeks
  any urgent or unscheduled visit to a clinician for worsening asthma symptoms during the 3 weeks after the index ED visit

CONTACTS AND LOCATIONS:
Locations (1):
- MetroHealth, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified information that allows replication of the main results